CLINICAL TRIAL: NCT06581172
Title: Significance of Disseminated Intravascular Coagulation Score in Mortality for Children With Shock
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nora Abdel Harith Amin, 71515,Assiut, Assiut University
Other Study IDs: DIC
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Shock, Septic
Keywords: DIC score
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: D_dimer — DIC score including FDPs,D_dimer

SUMMARY:
Evaluates whether the DIC score, as defined according to the International Society of Thrombosis and Hemostasis guidelines is associated with mortality in Children with shock and DIC

DETAILED DESCRIPTION:
Disseminated intravascular coagulation (DIC) is an acquired syndrome characterized by excessive systemic activation of coagulation, resulting in both hemorrhage and thrombosis. DIC can progress rapidly into lifethreatening multiorgan failure. Under normal hemostatic conditions, clot formation and resolution are tightly regulated. In DIC, dysregulated activation of the coagulation system results in a consumptive coagulopathy and microvascular thrombosis. DIC is always a secondary process caused by a variety of underlying disorders (eg, sepsis, trauma, or malignancy), which can cause endothelial tissue damage and procoagulant exposure .

This activates the coagulation cascade, which promotes fibrin production and deposition and consumption of clotting factors. The subsequent consumption of coagulation factors and platelets, inhibition of natural anticoagulants and fibrinolysis, and fibrin deposition result in the clinical picture of DIC: a bleeding diathesis accompanied by microvascular thrombosis that often leads to end-organ damage . The International Society of Thrombosis and Hemostasis and the Japanese Association for Acute Medicine scoring systems are useful for detection of the DIC in critically ill pediatric patients . The overall incidence of DIC to be 1.2%, using a scoring system comprised of etiologic factors, clinical features, platelet count, prothrombin time, fibrinogen, and fibrin degradation products (FDPs) . The DIC score, easily computed in real-time at the bedside with routine laboratory values, is associated with mortality for children with sepsis andshock.

Diagnosis of DIC through test of the D-dimer. Accordingly, testing for Ddimer or FDPs may be helpful for evulating relationship between DIC score and mortality rate among children with shock .

ELIGIBILITY:
Inclusion Criteria:

* All Children with shock and DIC will developed during the period from 1-1-2025 to 31-12-2025

Exclusion Criteria:

* Any shock not complicated with DIC

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with shock and DIC
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluates whether the DIC score, as defined according to the International Society of Thrombosis and Hemostasis guidelines is associated with mortality in Children with shock and DIC | Baseline
  Data of the patients will be collected in the
  form of:
  * Personal history (age, sex), demographics including residence.
  * Clinical history and examination including diagnoses, vital signs and signs of shock, cause of shock if detected.
  * Therapeutic history including the use of continuous vasoactive medications, volume of blood products transfused and the presence of mechanical ventilation
  Laboratory investigation:
  The four laboratory components of the DIC score were determined from
  1. Complete blood count (CBC).
  2. Prothrombin time (PT)
  3. Platelet count
  4. FDP titer Scoring systems The score was determined within the first 12 h of admission, at this time the patient was on the highest cumulative dose of these medications and used as a marker for hemodynamic instability. DIC scores were computed when all four-laboratory component
Scoring system | Baseline
  Component of the score 0 1 2 3 Max points possible
  Platelet count (/mm3 ) >100,000 100,000_51 ≤50,000 2 Fibrinogen (mg/dl) ≥100 <100 1 FDP titer (mg/ml) ≤5 6_40 >40 3 prolonged PT (s)<3 3_6 >6 2 Total score 8 All individual components are summed for a total of eight possible points. If d-dimer is used instead of FDP titer, then cutoff values for the DIC score are (0: ≤2 mg/l), (2: 2.1-8 mg/l) and (3: >8 mg/l)
  Interpretation of total score:
  ≥5 points positive for DIC <5 points: negative, but patients could still have "on_ overt DIC" which could evolve into Frank DIC .If there is ongoing concern for DIC, Coagulation labs may be repeated in 12_24 hours.

SECONDARY OUTCOMES:
Sample size | Baseline
  Eighty (80) children with shock will be included in this study during the period from 1-1-2025 to 31-12-2025. Sample size was calculated by Open Epi Info version (3) according to previous study conducted by Robinder., et al (2008), by comparing two related means using confidence level 85%.

REFERENCES:
- [Background] Chanthong S, Choed-Amphai C, Manowong S, Tuntivate P, Tansriratanawong S, Makonkawkeyoon K, Natesirinilkul R. Rotational Thromboelastometry and Clot Waveform Analysis as Point-of-Care Tests for Diagnosis of Disseminated Intravascular Coagulation in Critically Ill Children in Thailand. Pediatr Crit Care Med. 2024 May 1;25(5):e221-e231. doi: 10.1097/PCC.0000000000003452. Epub 2024 Feb 1. PMID 38299935
- [Background] Infante, J. B., Esteves, G. V., Raposo, J., & de Lacerda, J. F. (2024)
- [Background] Kim, T. W., Ko, R. E., Choi, K. H., Chung, C. R., Cho, Y. H., & Yang, J. H. (2024)
- [Background] Zafar A, Naeem F, Khalid MZ, Awan S, Riaz MM, Mahmood SBZ. Comparison of five different disseminated intravascular coagulation criteria in predicting mortality in patients with sepsis. PLoS One. 2024 Mar 7;19(3):e0295050. doi: 10.1371/journal.pone.0295050. eCollection 2024. PMID 38452037
- [Background] Rashad, A. B., Habib, M. S., Saleh, N. Y., & Abo El Fotoh, W. M. (2023)
- [Background] Songthawee N, Chavananon S, Sripornsawan P, McNeil E, Chotsampancharoen T. Prevalence and risk factors of disseminated intravascular coagulation in childhood acute lymphoblastic leukemia. Pediatr Res. 2023 Aug;94(2):588-593. doi: 10.1038/s41390-023-02475-8. Epub 2023 Jan 20. PMID 36670158
- [Background] Zhang, R., Huang, H., Lu, S., Chen, J., Pi, D., Dang, H., ... & Fu, Y. Q. (2024).
- [Background] Park, S. J., Oh, S. H., & Jhang, W. K. (2023, November).